CLINICAL TRIAL: NCT04208230
Title: Progression and Etiology of Cortical Porosity in Diabetic Bone Disease
Acronym: PREPT2D
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: iRIS 16-20196
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be frozen for future batch analysis of 1.25(OH)2D, sclerostin, the fat-secreted hormones (adipokines), adiponectin and leptin, estradiol, angiogenesis markers vascular endothelial growth factor (VEGF), angiopoietin-1 and antagonist ang-2, and the bone turnover markers C-terminal cross-linking telopeptide of type I collagen (CTX; bone resorption), total aminoterminal propeptide of type I collagen (PINP; bone formation), and bone-specific alkaline phosphatase (BAP; bone formation). Serum and urine will be stored for possible future analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects diagnosed with type 2 diabetes mellitus: Subjects with type 2 diabetes defined as those with (1) history and diagnosis of T2D and pharmacologic treatment for a minimum of 3 years OR (2) history and diagnosis of T2D with documented HgbA1C of 6.5 or higher for a minimum of 3 years if they are not under pharmacologic treatment (i.e., diet-controlled)
  Interventions: Device: XtremeCT
- Control: Non-diabetic control group. These subjects must not have pre-diabetes.
  Interventions: Device: XtremeCT

INTERVENTIONS:
Device: XtremeCT — HRpQCT technology provides information on bone microarchitecture, bone density and bone strength by measuring the cortical and trabecular bone structures with improved spatial resolution and defining the surfaces in three-dimensional manner.
  Other Names: High-resolution peripheral quantitative computed tomography (HRpQCT)

SUMMARY:
Type 2 diabetes is associated with increased cortical bone porosity and increased fracture risk. The goal of this proposed study is to understand the longitudinal evolution of cortical bone porosity and to investigate the underlying biological processes that drive increased cortical porosity and fracture risk in the setting of diabetes. The investigators will apply novel techniques for in vivo imaging of cortical pores to patients with type 2 diabetes and controls in a longitudinal prospective study. This work will establish the longitudinal progression of cortical porosity and determine whether pore content can serve as a predictor of future cortical degradation and bone fragility.

DETAILED DESCRIPTION:
The overall goal of this proposed study is to investigate the underlying biological processes that drive increased cortical porosity in the setting of Type 2 Diabetes and to understand the longitudinal evolution of human diabetic bone disease with a special focus on cortical porosity. The investigators propose the first longitudinal study of pore progression in T2D patients, which will be performed using a novel combined high-resolution peripheral quantitative computed tomography (HR-pQCT) and contrast enhanced magnetic resonance (CE MR) imaging approach. The investigators will use novel image analysis approaches to characterize pore content and spatial distribution of porosity within the cortex, and micro finite element (μFE) analysis to quantify biomechanical impact of porosity.

Bone quality deficits underlying increased fragility in T2D are not fully understood. At the tissue level, research evaluating deficits in material properties and fracture resistance is ongoing. At the structural level, increased cortical porosity is a clearly established deficit in bone quality in T2D. Porosity is a major determinant of strength, stiffness, and fracture toughness of cortical tissue, and therefore represents an important target for the prevention or reversal of T2D-associated skeletal fragility.

The mechanisms driving increased cortical porosity in T2D are unknown. To develop treatments specifically targeted at the prevention or reversal of pathological porosity, the investigators must understand the biological drivers of porosity. Today these biological drivers are unknown. Within the compact cortex, formation of large cortical pores has been attributed to clustering of osteons and merging of Haversian canals. At the endocortical border, 'trabecularization' or marrow space expansion is hypothesized to drive observed increases in cortical porosity. Multiple mechanisms of pore space expansion likely are at play in diabetic bone disease.

Increased marrow adiposity and compromised microvascular health are recognized aspects of T2D mellitus, and may be implicated in the development of pathological porosity. Studies investigating rodent models and humans have established the association of increased marrow fat with T2D. (BMI alone, in contrast, has not been shown to have an association with marrow fat.) Increased marrow fat - in turn - is associated with low Bone Mineral Density (BMD) and poor trabecular microstructure. The investigators have also documented that increased marrow fat is associated with vertebral fracture, independent of BMD. The historic concept of marrow fat as merely a passive filler has been superseded by an appreciation for this fat depot as a dynamic player in bone quality. To date this link has been studied primarily in terms of trabecular bone microstructure; the investigators propose that it could be a player in cortical bone microstructure as well. Microvascular complications of T2D are among the most serious manifestations of the disease. In advanced disease, neovascularization through the process of angiogenesis leads to progression of retinopathy and nephropathy. Recent work has suggested that microvascular pathology also affects trabecular bone quality in diabetes. In cortical bone, where the majority of porosity contains blood vessels, neovascularization necessitates removal of bone tissue. Therefore the investigators hypothesize that microvascular pathology may be influencing cortical microstructural changes in T2D.

Content of pathological pore space may indicate drivers of pore space expansion, and lead to strategies for predicting and preventing porosity-related fractures. Characterization of pore content may indicate pore space enlargement by expansion of the marrow cavity, expansion of the vascular network, or both. If the investigators discover that altered marrow distribution or composition is associated with increased porosity in T2D, this suggests that expansion of the marrow cavity may be contributing to pathological porosity. In this case the investigators would direct future efforts towards the emerging topic of fat-bone interactions, specifically: 1) the balance between osteoblast and adipocyte differentiation occurring from a common multipotent precursor; and 2) the action of adipokines on bone remodeling. If the investigators determine that altered vessel distribution or microvascular health is associated with increased porosity in T2D, this suggests that the vascular network may be contributing to pathological porosity. In this case the investigators would direct future research toward the interaction between the vascular system and cortical bone remodeling. The vascular system is known to influence bone remodeling through vasoactive substances released by endothelial cells. In the context of disuse, for example, bone loss is associated with increased vascularity and hyperemia, achieved by the release of vasoactive substances by endothelial cells. As the investigators look at these possible mechanisms of increased cortical porosity, appropriate treatment strategies will be clarified. Specifically, increased porosity related to fat metabolism might indicate interventions focused on directing mesenchymal stem cell differentiation towards osteoblastogenesis or regulating adipokine action on bone remodeling. Alternatively, increased porosity due to microvascular damage might indicate modulation of vasoregulators or anti-angiogenic therapy as used to combat neovascularization and bone erosion in rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female and/or male
* 50-70 years old
* Body mass index (BMI) of 18-40
* Subjects with bone mineral density of: 0 ≥ T-score > -2.5
* Additional requirement for type II diabetes patients:

  * Patients has a history of type II diabetes, as defined by the American Diabetes Association for more than 3 years. Patients must either have a documented HbA1C of 6.5 or higher for 3 or more years if they are not undergoing pharmacological treatment (diet controlled), or must have been receiving pharmacological treatment for the past 3 years.

Exclusion Criteria:

* Perimenopausal women, defined as last menses within previous 3 years
* History of metabolic bone disease other than post-menopausal bone loss. Persons with the following diseases: chronic gastrointestinal disease (including inflammatory bowel disease, celiac disease, or other malabsorptive disease including short-gut syndrome), renal or hepatic impairment (known cirrhosis or if transaminase levels 3 times the upper limit of normal)
* Current alcohol consumption (>3 alcohol drinks/day), current illicit drug use.
* Use of medications known to impact bone and mineral metabolism, including use of a bisphosphonate or teriparatide in the last year or for >12 months ever, current calcitonin, prednisone > 5mg daily or the equivalent glucocorticoid for > 10 days in the last 3 months, current thiazolidinedione (TZD), thyroid hormone replacement with current thyroid stimulating hormone < 0.1 miu/L. Patients undergoing hormone/testosterone replacement will NOT be excluded meaning they can be enrolled)
* Trauma or surgery near radius or tibia imaging sites
* An episode of immobilization lasting longer than 1 week in the previous 6 months
* Estimated Glomerular Filtration Rate (eGFR)< 50 mL/min/1.73 m2 (baseline) or < 40 (follow-up). The investigators will require eGFR ≥ 50 at baseline in an effort to avoid the possibility of an enrolled subject dropping below the established safety level of 40 at follow-up. This was determined knowing that eGFR can decline at a rate of approximately 4.0 per year in diabetics (much lower in non-diabetics).
* Conditions excluded by x-ray or MRI safety guidelines
* Body mass index greater than 40 as these subjects will be too large to fit into the gantry of the MR scanner or exceed weight limitations of the MR table

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes will be recruited from primary care clinics all over San Francisco;
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Amount of fat within cortical pores at the distal tibia at baseline | Baseline
  The investigators will apply a combined HR-pQCT and MR pore content characterization technique to quantify the amount of fat within cortical pores at the distal tibia in T2D subjects and matched controls.
Amount of vessels within cortical pores at the distal tibia at baseline. | Baseline
  The investigators will apply a combined HRpQCT and MR pore content characterization technique to quantify the proportion of cortical pores containing vessels at the distal tibia at baseline in T2D subjects and matched controls. .
Association between Type 2 diabetes status and marrow fat at the distal tibia | Baseline and 24 months
  Cortical porosity at the distal tibia will be assessed by HRpQCT at baseline and 24 months in T2D subjects and matched controls.

CONTACTS AND LOCATIONS:
Overall Officials: Galateia Kazakia, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No